CLINICAL TRIAL: NCT01825512
Title: Multicentre, Randomised, Open Label, Non-inferiority Trial to Evaluate the Efficacy and Safety of Deferiprone Compared to Deferasirox in Patients Aged From 1 Month to Less Than 18 Years Affected by Transfusion Dependent Haemoglobinopathies
Brief Title: Efficacy/Safety Study of Deferiprone Compared to Deferasirox in Paediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Consorzio per Valutazioni Biologiche e Farmacologiche (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEEP-2
Record Dates: First submitted 2013-04-03; First posted 2013-04-05 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2017-10

CONDITIONS: Chronic Iron Overload
Keywords: chronic iron overload; hereditary haemoglobinopathy; beta thalassaemia major; chelating agents; deferiprone; deferasirox; children; paediatrics
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferiprone; Isoflurophate; Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferiprone (Experimental): 75-100 mg/kg/day seven days per week
  Interventions: Drug: Deferiprone
- Deferasirox (Active Comparator): 20 to 40 mg/kg/day seven days per week
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferiprone — Deferiprone 80 mg/mL oral solution
  Other Names: DFP
  Arms: Deferiprone
Drug: Deferasirox — Deferasirox is used at the following dosage strengths: 125 mg, 250 mg and 500 mg
  Other Names: DFX; ATC Code:V03AC03
  Arms: Deferasirox

SUMMARY:
Multicentre, randomised, open label, non-inferiority active-controlled trial to evaluate efficacy and safety of a 12-months treatment with deferiprone (DFP) at dose of 75-100 mg/kg/day versus deferasirox (DFX) at dose of 20-40 mg/kg/day in paediatric patients (1 month < 18 years old) affected by hereditary haemoglobinopathies and requiring frequent transfusions and chelation.

DETAILED DESCRIPTION:
Haemoglobinopathies are a group of inherited disorders characterized by structural variations of the haemoglobin molecule. Most of the patients affected require for survival chronic red blood cells transfusions to overcome ineffective erythropoiesis. Unfortunately, all chronically transfused patients become clinically iron overloaded as there is no physiological mechanism for the removal of iron from the body. The pathologic changes and clinical manifestations associated to chronic iron overload are common among all transfusional iron-overload patients, albeit best documented in patients with beta-thalassemia major. The recommended treatment consists in regular blood transfusions combined with chelating therapy to remove the harmful iron accumulation in the body.

Currently, in the clinical practice particularly in children and adolescents, the criteria leading to the choice of the chelating agent include also the adherence to therapy, thus favouring the use of oral chelators (Ceci A et al., 2011) DFP (Deferiprone) was the first oral chelator authorised in Europe in 1999 as second line treatment for the treatment of iron overload in patients with thalassaemia major when DFO (Deferoxamine) is contraindicated or inadequate. However, despite a wide experience of DFP with iron overloaded (specifically thalassaemic )patients, limited data are available for younger children. For this reason the need for additional data in younger children is expressively included in the 2009 PDCO (Paediatric Committee) Priority List.

The purpose of this study is to assess the non-inferiority of DFP compared to DFX (deferasirox)in paediatric patients affected by hereditary haemoglobinopathies requiring chronic transfusions and chelation. Non inferiority will be established in terms of percentage of patients successfully chelated, as assessed by serum ferritin levels (in all patients) and cardiac MRI T2* (in patients above 10 years of age able to have an MRI scan without sedation).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged from 1 month up to less than 18 years at the time of enrolment
* Patients affected by any hereditary haemoglobinopathy requiring chronic transfusion therapy and chelation, including but not limited to thalassemia syndromes and sickle cell disease
* Patients on current treatment with deferoxamine (DFO) or DFX or DFP in a chronic transfusion program receiving at least 150 mL/kg/year of packed red blood cells (corresponding approximately to 12 transfusions);
* For patients naïve to chelation treatment: patients that have received at least 150 mL/kg of packed red blood cells (corresponding to approximately 12 transfusions) in a chronic transfusion program and with serum ferritin levels ≥ 800 ng/mL;
* Until availability of results from the PK Study (Study DEEP-1, EudraCT n. 2012-000658-67) for patients aged from 1 month to less than 6 years: known intolerance or contraindication to DFO;
* Written informed consent and patient's informed assent, relating to his/her comprehension abilities and level of maturity

Exclusion Criteria:

* Patients with intolerance or known contraindication to either DFP or DFX
* Patients receiving DFX at a dose > 40 mg/kg/day or DFP at a dose > 100 mg/kg/day at screening
* Platelet count <100.000/mm3 during the run-in phase
* Absolute neutrophils count <1.500/mm3 during the run-in phase
* Hb levels lower than 8g/dL during the run-in phase
* Evidence of abnormal liver function
* Iron overload from causes other than transfusional haemosiderosis
* Severe heart dysfunction secondary to iron overload
* Serum creatinine level > ULN (Upper Limit of Normal) for age during the run-in phase
* History of significant medical or psychiatric disorder
* The patient has received another investigational drug within 30 days prior to this clinical trial
* Fever and other signs/symptoms of infection in the 10 days before baseline assessment
* Concomitant use of trivalent cation-dependent medicinal products such as aluminium-based antacids
* Positive test for β-HCG (Human chorionic gonadotropin) and lactating female patients

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 435 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donato Bonifazi, Dr, Study Director — Consorzio per Valutazioni Biologiche e Farmacologiche; Aurelio Maggio, MD, Principal Investigator — Ospedali Riuniti Villa Sofia-Cervello
Locations (22):
- Albania (2):
  - Hospital 'Ihsan Çabej', Lushnjë
  - Qendra Spitalore Universitare "Nene Tereza" Tirane, Tirana
- Department of Medical and Public health Services of the Ministry of Health, Nicosia, Cyprus
- Egypt (3):
  - Alexandria University Hospital - Faculty of Medicine, Alexandria
  - Cairo University Faculty of Medicine, Cairo
  - Zagazig University Hospitals, Zagazig
- National And Kapodistrian University of Athens, Athens, Greece
- Italy (12):
  - Centro di Thalassemia, Ospedale Civile di Lentini, Lentini, SR
  - Università di Bari - Facoltà di Medicina, Bari
  - ASL Cagliari Ospedale Regionale per le Microcitemie, Cagliari
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - Presidio Ospedaliero "Annunziata", Centro di Studi della Microcitemia, Cosenza
  - A.O.Universitaria Meyer, Florence
  - Clinica Pediatrica Policlinico di Modena, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "Antonio Cardarelli", Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - U.O.C. Ematologia - Emoglobinopatie, Ospedale G. Di Cristina, Palermo
  - Clinica Pediatrica Università - ASL 1 D.H per Talassemia, Sassari
- Centre National de Greffe de Moelle Osseuse Tunis, Tunis, Tunisia
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Queen's Hospital, Romford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giannuzzi V, Felisi M, Bonifazi D, Devlieger H, Papanikolaou G, Ragab L, Fattoum S, Tempesta B, Reggiardo G, Ceci A. Ethical and procedural issues for applying researcher-driven multi-national paediatric clinical trials in and outside the European Union: the challenging experience of the DEEP project. BMC Med Ethics. 2021 Apr 29;22(1):49. doi: 10.1186/s12910-021-00618-2. PMID 33926431
- [Derived] Maggio A, Kattamis A, Felisi M, Reggiardo G, El-Beshlawy A, Bejaoui M, Sherief L, Christou S, Cosmi C, Della Pasqua O, Del Vecchio GC, Filosa A, Cuccia L, Hassab H, Kreka M, Origa R, Putti MC, Spino M, Telfer P, Tempesta B, Vitrano A, Tsang YC, Zaka A, Tricta F, Bonifazi D, Ceci A. Evaluation of the efficacy and safety of deferiprone compared with deferasirox in paediatric patients with transfusion-dependent haemoglobinopathies (DEEP-2): a multicentre, randomised, open-label, non-inferiority, phase 3 trial. Lancet Haematol. 2020 Jun;7(6):e469-e478. doi: 10.1016/S2352-3026(20)30100-9. PMID 32470438
- See also: official project website — http://www.deepproject.eu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed consent was collected for 435 patients that were enrolled in the study, however 42 of them were excluded from the study for the following reasons: 17 did not meet inclusion criteria, 5 withdrew the consent and 20 were lost to follow-up.
Period: Baseline
Arm/Group | Deferiprone | Deferasirox
Started | 194 | 199
Completed | 193 | 197
Not Completed | 1 | 2
Period: Treatment
Arm/Group | Deferiprone | Deferasirox
Started | 193 | 197
Completed | 140 | 170
Not Completed | 53 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferiprone | Deferasirox | Total
Number analyzed (Participants) | 193 | 197 | 390
Age, Customized [Number; unit: participants]
  <6 years | 59 | 58 | 117
  > or equal to 6 years and <10 years | 47 | 47 | 94
  > or equal to 10 years | 87 | 92 | 179
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 93 | 173
  Male | 113 | 104 | 217
Race/Ethnicity, Customized [Number; unit: participants]
  Europe | 56 | 56 | 112
  North Africa | 121 | 122 | 243
  Rest of Africa | 6 | 5 | 11
  Asia | 0 | 1 | 1
  North America | 0 | 0 | 0
  Latin America | 0 | 0 | 0
  Other | 5 | 6 | 11
  Missing | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 12 | 23
  Italy | 30 | 28 | 58
  Tunisia | 28 | 28 | 56
  Egypt | 96 | 99 | 197
  Albania | 19 | 20 | 39
  Greece | 5 | 6 | 11
  Cyprus | 4 | 4 | 8
Ferritin level [Mean (Standard Deviation); unit: ng/ml] — Population: The difference is due to missing data at baseline
  ng/ml
    number analyzed (Participants) | 163 | 173 | 336
    (all) | 2756 (2175) | 2989 (2409) | 2876 (2298)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successfully Chelated Patients
Description: Percentage of successfully chelated patients is assessed by serum ferritin levels (in all patients) and cardiac MRI T2* (in patients above 10 years of age able to perform an MRI scan without sedation)
Time Frame: at baseline and after 12 months
Population: Per-protocol population 1 (PP1): number of patients for whom the primary composite efficacy endpoint data were available at baseline and after 1 year of treatment (271 subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone | Deferasirox
Number analyzed (Participants) | 125 | 146
Participants | 69 | 80
Statistical Analysis 1: Comparison: Deferiprone vs Deferasirox; Test type: Non-Inferiority — Deferiprone was declared non inferior to Deferasirox if the lower limit of the 95% confidence interval for the difference in the proportion of successful chelation in the two groups is above -12.5%; Treatment success rate = -12.5, 95% CI 1-sided [lower limit -12.5]

2. Secondary Outcome: Liver MRI
Description: Change in liver iron concentration (measured using liver MRI), assessed as difference between value at 12 months minus value at baseline.
Time Frame: at baseline and after 12 months
Population: Per-protocol population 3 (PP3): number of patients for whom liver iron concentration were available at baseline and after 1 year of treatment (106 subjects)
Measure: Mean (Standard Error); unit: mg/g
Arm/Group | Deferiprone | Deferasirox
Number analyzed (Participants) | 46 | 60
mg/g | -0.848 (0.887) | -2.975 (0.776)
Statistical Analysis 1: Comparison: Deferiprone vs Deferasirox; Test type: Other — GLM model; p = 0.074, ANCOVA; Mean Difference (Final Values) = 2.128, 95% CI 2-sided [-0.213 to 4.468], Standard Error of Mean 1.18

3. Secondary Outcome: Cardiac MRI T2*
Description: Change in cardiac iron concentration (measured using cardiac MRI T2*), assessed as difference between value at 12 months minus value at baseline. MRI T2* is a non-invasive method based on gradient echo (GRE) sequences, where T2* represents the spin-spin relaxation times, measured in milliseconds. The faster the curve decreases (ie, the smaller T2*), the greater amount of iron is in the tissue. Treatment success was assessed as follows: if baseline cardiac T2* was less than 20 ms, an increase of 10% or more after 1 year of treatment was defined as treatment success; if baseline cardiac T2* was more than 20 ms, any increase or a decrease of less than 10% after 1 year of treatment was defined as treatment success.
Time Frame: at baseline and after 12 months
Population: Per-protocol population 3 (PP3): number of patients for whom cardiac T2* concentration were available at baseline and after 1 year of treatment (108 subjects)
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | Deferiprone | Deferasirox
Number analyzed (Participants) | 49 | 59
milliseconds (ms) | 0.488 (1.284) | 1.121 (1.169)
Statistical Analysis 1: Comparison: Deferiprone vs Deferasirox; Test type: Other — GLM Analysis; p = 0.717, ANCOVA; Mean Difference (Final Values) = -0.633, 95% CI 2-sided [-4.085 to 2.819], Standard Error of Mean 1.741

4. Secondary Outcome: Ferritin Level
Description: Change in serum ferritin level, assessed as difference between value at 12 months minus value at baseline.
Time Frame: at baseline and after 12 months
Population: Per-protocol population 2 (PP2): number of patients for whom the per-protocol centralised serum ferritin concentration data were available at baseline and after 1 year of treatment (303 subjects, this population was larger than PP1 because PP2 included patients who did not have cardiac T2* data)
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Deferiprone | Deferasirox
Number analyzed (Participants) | 137 | 166
ng/mL | -397.583 (121.794) | -398.184 (110.619)
Statistical Analysis 1: Comparison: Deferiprone vs Deferasirox; Test type: Non-Inferiority — Non inferiority of Deferiprone to Deferasirox is tested considering a non-inferiority margin of 400 ng/mL; p = 0.997, GLM; Mean Difference (Final Values) = 0.601, 95% CI 2-sided [-323.580 to 324.781], Standard Error of Mean 164.734

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year for subject
Arm/Group | Deferiprone | Deferasirox
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/197
Serious Adverse Events (participants affected / at risk) | 13/193 | 14/197
Other Adverse Events (participants affected / at risk) | 152/193 | 89/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=193) | Deferasirox (N=197)
testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — testicular injury
splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — splenectomy
agranulocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — agranulocytosis
neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — neutropenia
sickle cell anaemia with crisis subjects affected/exposed (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — sickle cell anaemia with crisis subjects affected/exposed
seizure (Nervous system disorders) | 1 (1) | 0 (0) — seizure
pyrexia (General disorders) | 1 (1) | 1 (1) — pyrexia
chest pain (General disorders) | 0 (0) | 2 (2) — chest pain
gait disturbance (General disorders) | 0 (0) | 1 (1) — gait disturbance
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) — diarrhoea
hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 1 (1) — hypertransaminasaemia
acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) — acute kidney injury
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — pain in extremity
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) — gastroenteritis
meningitis meningococcal (Infections and infestations) | 0 (0) | 1 (1) — meningitis meningococcal
herpangina (Infections and infestations) | 0 (0) | 1 (1) — herpangina
pneumonia (Infections and infestations) | 2 (2) | 1 (1) — pneumonia
subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) — subcutaneous abscess
urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) — urinary tract infection
herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) — herpes virus infection
impetigo (Infections and infestations) | 0 (0) | 1 (1) — impetigo
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) — upper respiratory tract infection
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=193) | Deferasirox (N=197)
cough (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 16 (25) — cough
neutropenia (Blood and lymphatic system disorders) | 18 (26) | 11 (15)
pyrexia (General disorders) | 28 (40) | 32 (56)
abdominal pain (General disorders) | 20 (24) | 8 (9)
vomiting (General disorders) | 33 (42) | 8 (10)
arthralgia (Musculoskeletal and connective tissue disorders) | 23 (28) | 5 (5)
pharyngitis (Infections and infestations) | 15 (18) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT01825512/Prot_SAP_000.pdf